CLINICAL TRIAL: NCT03950596
Title: Macroscopic and Molecular Changes in Knee Muscular-tendon Unit in Response to Acute Resistant Load
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HYMC-58-16
Record Dates: First submitted 2019-05-01; First posted 2019-05-15 (Actual); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Quadriceps Muscle
MeSH Terms: interventions — DNA; Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- One acute resistance load exercise (Active Comparator): One hundred volunteers will participate in one acute resistance load exercises to their quadriceps
  Interventions: Other: Acute resistant load exercises; Behavioral: Background Questionnaire; Other: Pain Questionnaire; Genetic: DNA and RNA test; Diagnostic Test: Ultrasound; Diagnostic Test: Percutaneous Needle Core Biopsy
- Three acute resistance load exercises (Active Comparator): One hundred volunteers will participate in three acute resistance load exercises to their quadriceps
  Interventions: Other: Acute resistant load exercises; Behavioral: Background Questionnaire; Other: Pain Questionnaire; Genetic: DNA and RNA test; Diagnostic Test: Ultrasound; Diagnostic Test: Percutaneous Needle Core Biopsy
- Control Group (Active Comparator): One hundred volunteers will participate in study as a control group
  Interventions: Behavioral: Background Questionnaire; Other: Pain Questionnaire; Genetic: DNA and RNA test; Diagnostic Test: Ultrasound; Diagnostic Test: Percutaneous Needle Core Biopsy

INTERVENTIONS:
Other: Acute resistant load exercises — Leg bench and leg press acute resistant load exercises
  Leg-bench and leg-press acute resistant load exercises
  Arms: One acute resistance load exercise; Three acute resistance load exercises
Behavioral: Background Questionnaire — Background questionnaire will be filled out by participants
Other: Pain Questionnaire — Pain questionnaire regarding pain in the knee during previous 3 months
Genetic: DNA and RNA test — DNA and RNA tests will be sent to a genetic laboratory for analysis
Diagnostic Test: Ultrasound — Ultrasound of the knee joint and the quadriceps muscle and the pica tendon
Diagnostic Test: Percutaneous Needle Core Biopsy — Core Biopsy will be taken from the quadriceps femoris muscle

SUMMARY:
The aim of this study is to determine the influence of acute resistance exercises on anatomical and biological changes in the quadriceps muscle and tendons of the knee

ELIGIBILITY:
Inclusion Criteria:

* Non-professional athletes
* Pass heart/lung endurance tests
* Pass ergometrics testing

Exclusion Criteria:

* Have been injured
* Had physiotherapy for back or lower limbs in past 6 months
* Orthopedic surgery in lower limbs

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-05 (Estimated); Primary Completion 2020-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Genetic Changes in Knee Muscle and Tendon | One year
  Comparison of results of genetic testing both before and after interventions between the 3 groups
Ultrasound Changes in Knee Muscle and Tendon | One year
  Comparison of results of pre- and post ultrasound changes after interventions between the 3 groups
Biopsy Changes in Knee Muscle and Tendon | One year
  Comparison of changes in biopsies taken before and after interventions between the 3 groups

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel

IPD SHARING:
Plan to Share IPD: No